CLINICAL TRIAL: NCT06967636
Title: The Impact of Successful Quitting Smoking After the Intensive Gold Standard Programme (GSP) on Morbidity and Mortality Among Smokers With Severe Mental Disorders - A Nationwide Cohort Study From the Danish STOPbase
Brief Title: The Impact of Successful Quitting Smoking After Intensive Smoking Cessation Interventions on Morbidity and Mortality Among Smokers With Severe Mental Disorders - A Nationwide Cohort Study From the Danish Smoking Cessation Database
Status: Completed | Type: Observational
Sponsor: Parker Research Institute (Other)
Responsible Party: Principal Investigator, Sine Holst-Albrechtsen, MD, MSc, Parker Research Institute
Other Study IDs: 2000-54-0013; STOPbase (Registry Identifier: The STOPbase - The Danish smoking cessesation databse); NPR (Registry Identifier: NPR - The Danish National Patient Register); RCD (Registry Identifier: RCD - The Danish National Registry of Causes of Death)
Record Dates: First submitted 2025-05-05; First posted 2025-05-13 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Smoking Cessation, Mental Health Disorders, Inequality in Health Prevention
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
We evaluate intensive smoking cessation interventions (GSP) on morbidity and mortality in terms of assessing the impact among quitters and non-quitters with severe mental disorders (SMD)

ELIGIBILITY:
Inclusion Criteria:

* F20-F29, F30-F39, F60-F69, F10-F16, F18, F19
* Participation in the GSP in Denmark

Exclusion Criteria:

* Dual diagnosis (F00-F99 and a co-occurring substance-use disorder (F10-F16, F18, F19)
* < 18 years
* No consent to follow-up
* No baseline smoking status

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All participants >18 years with a severe mental disorder (SMD) undergoing the GSP in Denmark at local clinics with consent to follow up.
Sampling Method: Non-Probability Sample
Enrollment: 15863 (Actual)
Dates: Start 2006-01-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
All-cause morbidity | January 2006 to January 2020
  Days of hospital contact of all causes
All-cause mortality | January 2006 to January 2023
  Death from all causes